CLINICAL TRIAL: NCT07177833
Title: Title Fractioned CO2 Laser in the Treatment of Chronic Phase Peyronie's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240299-01H
Record Dates: First submitted 2025-08-26; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Peyronies Disease
Keywords: Peyronies disease
MeSH Terms: conditions — Penile Induration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fractional CO2 laser therapy group (Experimental): Patients will receive three treatments with fractional CO2 laser to identified Peyronie's plaque tissue
  Interventions: Device: Fractional CO2 laser
- Sham control group (Sham Comparator): Patients will receive sham treatment with non-invasive treatment mimicking CO2 laser therapy
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Device: Fractional CO2 laser — Fractional CO2 Laser Therapy is an extra-dermal (applied to the surface of the skin) and non-invasive treatment that involves the use of lasers to destroy and reduce abnormal collagen in scarred tissue.
  Arms: Fractional CO2 laser therapy group
Other: Sham (No Treatment) — Patients will undergo a treatment with a vibratory device capable of mimicking fractional CO2 laser therapy
  Arms: Sham control group

SUMMARY:
Peyronie's Disease (PD) is a fibrosing disorder of the penis where scar tissue (composed of excessive and disorganized collagen) known as a "plaque," forms along the shaft of the penis. This plaque can lead to permanent penile deformity (curvature, narrowing, indentation, hinging), loss of penile length, erectile dysfunction, and pain during intercourse. Research has shown PD to negatively impact the quality of life and cause significant psychosocial distress for many men.

At present, available medical and surgical treatment modalities for PD have limitations. Intralesional collagenase clostridium histolyticum (CCh) is approved for the reduction of penile curvature in PD, however, its use is restricted to the United States market. Other medical therapies including intralesional verapamil and interferon injections have inconsistent and modest effects while, invasive surgical management with plication or grafting can result in erectile dysfunction, penile length shortening, penile sensory changes, and harvest site complications.

Fractional CO2 Laser Therapy is an extra-dermal (applied to the surface of the skin) and non-invasive treatment that involves the use of lasers to destroy and reduce abnormal collagen in scarred tissue. Most recently, it has been used in a pilot clinical trial investigating its use in the management of PD. All men in this study safely experienced reduction in their penile curvature.

This will be a phase 1 clinical trial evaluating the safety and feasibility of using a fractional CO2 laser in the management of chronic phase PD. Enrolled study participants will undergo an initial clinical assessment of their PD which involves penile measurements at flaccid and erect states, a curvature assessment with duplex ultrasound, and will be asked to complete the International Index of Erectile Function Questionnaire (IIEF-5), and Peyronie's Disease Questionnaire (PDQ). They will then undergo 3 laser therapy sessions at 6 week intervals and will have a short and long-term follow-up of 24 and 52 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Men 18 or older. For heterosexual men it is required they be in a stable relationship with a female spouse/partner for at least 3 months and willing to have vaginal intercourse for purposes of properly filling out the validated PD Questionnaire.
2. Diagnosis of PD for at least 12 months with evidence of stable disease as determined by the investigator (i.e. no change in penile curve for at least 6 months and absence of pain).
3. Penile curvature of 30º-90º in the dorsal, lateral, or dorsal/lateral plane (must be possible to delineate the single plane of maximal curvature for evaluation)
4. Signed informed REB-approved consent agreement; signed authorization form to allow disclosure of protected information.
5. Ability to read, complete, and understand the various rating instruments in English.

Exclusion Criteria:

1. Penile curvature of <30º or >90º
2. Any conditions affecting the penis such as a chordee in the presence or absence of hypospadias; thrombosis of the dorsal penile artery; infiltration by a benign or malignant mass or an infectious agent; ventral curvature from any cause; presence of an active sexually transmitted disease.
3. Failure to achieve a sufficient 8/10 erection (after prostaglandin E or Trimix administration), in the opinion of the investigator, to accurately measure the penile deformity.
4. Calcified plaque as evident by appropriate radiographic evaluation, i.e., penile ultrasound that would prevent treatment with Fractional CO2 Laser
5. Isolated hourglass deformity of the penis without curvature
6. Treatment or plans to undergo treatment for PD, including but not limited to any previous surgery, oral/topical agents within 3 months, intralesional medical therapies within 3 months, extracorporeal shock wave therapy within 6 months, or use of mechanical devices within 2 weeks before the start of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety of fractional CO2 laser therapy application to Peyronie's plaque tissue | 52 week follow up period
  Proportion of participants experiencing treatment-related adverse events (AEs) and serious adverse events (SAEs) following three sessions of fractional CO₂ laser therapy for Peyronie's disease. Safety will be assessed through patient self-reports, clinical evaluations at each visit, and documentation in adverse event logs.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Witherspoon, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No